CLINICAL TRIAL: NCT02910635
Title: A Randomized, Placebo-Controlled, Four-Period Crossover, Study to Evaluate the Effect of Volanesorsen on the QTc Interval Using a Therapeutic and Supra-Therapeutic Dose Compared With Placebo in Healthy Volunteers: a Thorough QT Study
Brief Title: A Study to Evaluate the Effect of Volanesorsen on Cardiac Repolarization Conducted in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Collaborators: Akcea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: ISIS 304801-CS13
Record Dates: First submitted 2016-09-09; First posted 2016-09-22 (Estimated); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Abnormalities, Cardiovascular
Keywords: Thorough QTc, Therapeutic dose, supra therapeutic dose
MeSH Terms: conditions — Cardiovascular Abnormalities | interventions — ISIS 304801; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Volanesorsen, Intravenous (IV) (Experimental): 300 mg of volanesorsen (ISIS 304801) administered Intravenous (IV) single dose
  Interventions: Drug: Volanesorsen
- Volanesorsen, Subcutaneous (SQ) (Experimental): 300 mg of volanesorsen (ISIS 304801) administered Subcutaneous (SQ) single dose
  Interventions: Drug: Volanesorsen
- Moxifloxacin Hydrochloride (Active Comparator): Moxifloxacin Hydrochloride 400 mg tablet administered orally, Single Dose
  Interventions: Drug: Moxifloxacin
- Placebo Intravenous (IV) single dose (Placebo Comparator): Administered as normal saline (0.9% Sodium Chloride)
  Interventions: Drug: Placebo
- Placebo Subcutaneous (SC) single dose (Placebo Comparator): Administered as normal saline (0.9% Sodium Chloride)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Volanesorsen — ISIS 304801 is supplied as 200mg of volanesorsen with 1.0mL of solution per vial
  Arms: Volanesorsen, Intravenous (IV); Volanesorsen, Subcutaneous (SQ)
Drug: Moxifloxacin — Moxifloxacin Hydrochloride 400 mg tablet administered orally, Single Dose
  Arms: Moxifloxacin Hydrochloride
Drug: Placebo
  Arms: Placebo Intravenous (IV) single dose; Placebo Subcutaneous (SC) single dose

SUMMARY:
The primary objective of this study is to assess the corrected QT interval (QTc) effect of volanesorsen (ISIS 304801) administered as a 300 mg subcutaneous (SC) therapeutic and a 300 mg intravenous (IV; 2-hour infusion) supra-therapeutic dose relative to placebo in healthy adult male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Must have given written informed consent and be able to comply with all study requirements
* Males and females aged 18-55 at the time of informed consent
* Females must be non-pregnant and non-lactating surgically sterile, post-menopausal or if engaged in sexual relations of childbearing potential, using an acceptable contraceptive method
* Males must be surgically sterile, abstinent or using an acceptable contraceptive method
* The subject has a BMI of 19 to 32 kg/m^2 inclusive
* Consumption of nicotine or nicotine-containing products for at least 6 months before Screening

Exclusion Criteria:

* History of risk factors for Torsades de Pointes, unexplained syncope, known Long QT Syndrome, heart failure, myocardial infarction, angina, or clinical significant abnormal laboratory assessments including hypokalemia, hypocalcemia, hypercalcemia, or hypomagnesemia
* Abnormal screening ECG
* Use of concomitant medications unless authorized by the Sponsor Medical Monitor
* Known history of or positive test for human immunodeficiency virus (HIV), hepatitis C or chronic hepatitis B
* Treatment with another Study Drug, biological agent, or device within one-month of Screening
* Tests positive for drugs of abuse or cotinine
* Considered unsuitable for inclusion by the Principal Investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2016-09-19 (Actual); Primary Completion 2016-12-20 (Actual); Study Completion 2016-12-20 (Actual)

PRIMARY OUTCOMES:
Placebo corrected change from baseline in QTcF (corrected Frederica's CT Interval) | 24 Hours
  ECG monitoring up to 24 hours post dose

SECONDARY OUTCOMES:
Placebo corrected change from baseline heart rate (HR, PR and QRS) | 24 Hours
  ECG monitoring 24 hours post dose

OTHER OUTCOMES:
Volanesorse plasma pharmacokinetics (PK) | 0 to 24 hours
  Area under the plasma concentration time curve from time 0 to 24 hours (AUC 0-24h)

CONTACTS AND LOCATIONS:
Locations (1):
- Covance, Dallas, Texas, United States